CLINICAL TRIAL: NCT03903276
Title: Effects of Transcutaneous Electrical Nerve Stimulation in the Conventional Mode in Post-operative Lung Cancer Patients in a Reference Hospital in the Amazon Region
Brief Title: Effects of Transcutaneous Electrical Nerve Stimulation in Post-operative Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Collaborators: Universidade do Estado do Pará (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, Phd, Director of Human Movement Department, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90466098200
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Cancer, Lung
MeSH Terms: conditions — Lung Neoplasms | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): assessment of pain scale and functional capacity
- Experimental (Experimental): assessment of pain scale and functional capacity, TENS 30 minutes 3 sessions
  Interventions: Other: rehabilitation

INTERVENTIONS:
Other: rehabilitation — Tens
  Arms: Experimental

SUMMARY:
Among all cancers, lung cancer is the most common disease on the planet, accounting for 13% of the cases, and leading the number of deaths from malignant diseases. In Brazil, it is estimated that its incidence between 2018 and 2019 could be 18,704 new cases in men and 12,503,000 new cases in women. These data take into account an estimated risk of 18.16 new cases for 100,000 men and 11.81 for 100,000 women, respectively occupying the second and fourth most frequent cases of the disease according to gender .

Surgeries, however aggressive they may be, are one of the most viable alternatives for patients with PC, provided it is performed in the milder or early phase of the disease, since after such period this procedure may have a period degree greater than the other forms of treatment.

As a consequence, the injuries that the surgical procedure can cause to patients, pain is one of the most influential in the patient's quality of life. It can lead the individual to a marked state of disability both functional and psychological, thus being determinant for the suffering related to the disease, thus comprising its multifactorial character, involving physical, emotional, socio-cultural and environmental aspects .

For the control of pain, physiotherapy appears with features such as transcutaneous nerve electrostimulation, where its use for the suppression of pain has become quite feasible due mainly to the ease of its handling, to be noninvasive and to serve to reduce acute pain and chronic.

The use of conventional transcutaneous nerve electrostimulation to support the use of analgesics reduced the intensity of pain in patients of the second day of thoracotomy, but for a longer extension of their effects, it would take a longer time to apply the resource, something around 24 -48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Primary Lung Cancer; male over 18 years and less than 59 years old, in an immediate postoperative period in the ward of the Hospital thoracic clinic.
* Evaluation of pain through the visual analogue scale equal to or greater than moderate or intense.
* Percentage equal to or greater than 70% in all the items assessed by the Performance Status functional capacity scale.

Exclusion Criteria:

* Patients with immediate postoperative complications
* Unconscious or sedation patients
* Patients with invasive mechanical ventilation
* Patients who present lesions that make it difficult to handle and place electrodes.
* Patients who use pacemakers and metal plates.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Pain perception | post treatment in 3 days
  Visual analogue scale - EVA: consists of checking the intensity of pain in patients at the moment it is being evaluated. Such a tool consists of a line with the ends numbered from 0 to 10, and from 0 to 2 it is considered light pain; 3 to 7 moderate pain; and 8 to 10 severe pain
Functional capacity | post treatment in 3 days
  Functional capacity scale Performance Status- PS: aims to monitor the clinical evolution of a disease by joining the Karnofsky scale and the Zubrod or ECOG scale. Karnofsky's scale or index describes increasing levels of activities and independence of the individual stipulated values between 0 and 100, zero meaning no functionality or death and 100 representing the maximum degree of physical ability to perform activities. The Zubrod or ECOG scale quantified between 0 and 4, where 0 means 0 indicates that the individual is fully active for the performance of his activities and 4 assigning to the dead patient. Such scales are widely used for the evaluation of oncological patients, being somewhat complementary, therefore used together

CONTACTS AND LOCATIONS:
Overall Officials: Jadson Poça, graduated, Study Chair — Universidade do Estado do Pará
Locations (1):
- Universidade do Estado do Pará, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ainsworth L, Budelier K, Clinesmith M, Fiedler A, Landstrom R, Leeper BJ, Moeller L, Mutch S, O'Dell K, Ross J, Radhakrishnan R, Sluka KA. Transcutaneous electrical nerve stimulation (TENS) reduces chronic hyperalgesia induced by muscle inflammation. Pain. 2006 Jan;120(1-2):182-187. doi: 10.1016/j.pain.2005.10.030. Epub 2005 Dec 19. PMID 16360266
- [Result] Spiro SG, Gould MK, Colice GL; American College of Chest Physicians. Initial evaluation of the patient with lung cancer: symptoms, signs, laboratory tests, and paraneoplastic syndromes: ACCP evidenced-based clinical practice guidelines (2nd edition). Chest. 2007 Sep;132(3 Suppl):149S-160S. doi: 10.1378/chest.07-1358. PMID 17873166
- [Result] Hochberg U, Elgueta MF, Perez J. Interventional Analgesic Management of Lung Cancer Pain. Front Oncol. 2017 Feb 14;7:17. doi: 10.3389/fonc.2017.00017. eCollection 2017. PMID 28261561
- [Result] Rushton DN. Electrical stimulation in the treatment of pain. Disabil Rehabil. 2002 May 20;24(8):407-15. doi: 10.1080/09638280110108832. PMID 12033995